CLINICAL TRIAL: NCT06615869
Title: A Study to Evaluate the Pharmacokinetics and Definitive Bioequivalence of Molnupiravir Tablet Formulation Compared to the Molnupiravir Capsule Formulation in Healthy Adult Participants
Brief Title: A Study to Evaluate Molnupiravir Tablet Formulation Compared to the Molnupiravir Capsule Formulation in Healthy Adult Participants (MK-4482-011)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 4482-011; MK-4482-011 (Other: MSD)
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Healthy
MeSH Terms: interventions — molnupiravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Molnupiravir Treatment A (Experimental): Participants receive molnupiravir reference capsule.
  Interventions: Drug: Molnupiravir
- Molnupiravir Treatment B (Experimental): Participants receive molnupiravir Formulation 1.
  Interventions: Drug: Molnupiravir
- Molnupiravir Treatment C (Experimental): Participants receive molnupiravir Formulation 1 after a high-fat meal.
  Interventions: Drug: Molnupiravir
- Molnupiravir Treatment D (Experimental): Participants receive molnupiravir Formulation 2.
  Interventions: Drug: Molnupiravir

INTERVENTIONS:
Drug: Molnupiravir — Oral Administration.
  Other Names: MK-4482; MOV; LAGEVRIO; EIDD-2801

SUMMARY:
The goal of the study is to learn what happens to different forms of molnupiravir (MOV) medications in a healthy person's body over time when taken on an empty stomach or with food. Researchers will compare the amount of MOV in the healthy person's body over time when different forms of medications are given.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

- Has body mass index (BMI) ≥18 kg/m^2 and ≤32 kg/m^2.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* History of significant multiple and/or severe allergies (eg, food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (ie, systemic allergic reaction) to prescription or nonprescription drugs or food.
* Positive test(s) for Hepatitis B surface antigen (HBsAg), hepatitis C antibodies or Human immunodeficiency virus (HIV).
* History of a major surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of N-Hydroxycitidine (NHC) in plasma: Treatment A versus Treatment B | Pre-dose, and at designated timepoints up to 72 hours postdose
  AUC0-inf of NHC in plasma will be determined.
Area Under the Concentration-Time Curve From Time Zero to last measurable timepoint (AUC0-last) of NHC in plasma: Treatment A versus Treatment B | Pre-dose, and at designated timepoints up to 72 hours postdose
  AUC0-last of NHC in plasma will be determined.
Area Under the Concentration-Time Curve From Time Zero to 12 hours (AUC0-12) of (NHC) in plasma: Treatment A versus Treatment B | Pre-dose, and at designated timepoints up to 12 hours postdose
  AUC0-12 of NHC in plasma will be determined.
Maximum plasma concentration (Cmax) of NHC: Treatment A versus Treatment B | Pre-dose, and at designated timepoints up to 72 hours postdose
  Cmax of NHC in plasma will be determined.
Time to maximum plasma concentration (Tmax) of NHC: Treatment A versus Treatment B | Pre-dose, and at designated timepoints up to 72 hours postdose
  Tmax of NHC in plasma will be determined.
Apparent terminal half-life (t1/2) of NHC in plasma: Treatment A versus Treatment B | Pre-dose, and at designated timepoints up to 72 hours postdose
  t1/2 of NHC in plasma will be determined.
Apparent Clearance (CL/F) of NHC in plasma: Treatment A versus Treatment B | Pre-dose, and at designated timepoints up to 72 hours postdose
  CL/F of NHC in plasma will be determined.
Apparent volume of distribution during terminal phase (Vz/F) of NHC in plasma: Treatment A versus Treatment B | Pre-dose, and at designated timepoints up to 72 hours postdose
  Vz/F of NHC in plasma will be determined.

SECONDARY OUTCOMES:
AUC0-inf of NHC in plasma: Treatment B versus Treatment C | Pre-dose, and at designated timepoints up to 72 hours postdose
  AUC0-inf of NHC in plasma will be determined.
AUC0-last of NHC in plasma: Treatment B versus Treatment C | Pre-dose, and at designated timepoints up to 72 hours postdose
  AUC0-last of NHC in plasma will be determined.
AUC0-12 of NHC in plasma: Treatment B versus Treatment C | Pre-dose, and at designated timepoints up to 12 hours postdose
  AUC0-12 of NHC in plasma will be determined.
Cmax of NHC in plasma: Treatment B versus Treatment C | Pre-dose, and at designated timepoints up to 72 hours postdose
  Cmax of NHC in plasma will be determined.
Tmax of NHC in plasma: Treatment B versus Treatment C | Pre-dose, and at designated timepoints up to 72 hours postdose
  Tmax of NHC in plasma will be determined.
t1/2 of NHC in plasma: Treatment B versus Treatment C | Pre-dose, and at designated timepoints up to 72 hours postdose
  t1/2 of NHC in plasma will be determined.
CL/F of NHC in plasma: Treatment B versus Treatment C | Pre-dose, and at designated timepoints up to 72 hours postdose
  CL/F of NHC in plasma will be determined.
Vz/F of NHC in plasma: Treatment B versus Treatment C | Pre-dose, and at designated timepoints up to 72 hours postdose
  Vz/F of NHC in plasma will be determined.
AUC0-inf of NHC in plasma: Treatment D versus Treatment A | Pre-dose, and at designated timepoints up to 72 hours postdose
  AUC0-inf of NHC in plasma will be determined.
AUC0-last of NHC in plasma: Treatment D versus Treatment A | Pre-dose, and at designated timepoints up to 72 hours postdose
  AUC0-last of NHC in plasma will be determined.
AUC0-12 of NHC in plasma: Treatment D versus Treatment A | Pre-dose, and at designated timepoints up to 12 hours postdose
  AUC0-12 of NHC in plasma will be determined.
Cmax of NHC in plasma: Treatment D versus Treatment A | Pre-dose, and at designated timepoints up to 72 hours postdose
  Cmax of NHC in plasma will be determined.
Tmax of NHC in plasma: Treatment D versus Treatment A | Pre-dose, and at designated timepoints up to 72 hours postdose
  Tmax of NHC in plasma will be determined.
t1/2 of NHC in plasma: Treatment D versus Treatment A | Pre-dose, and at designated timepoints up to 72 hours postdose
  t1/2 of NHC in plasma will be determined.
CL/F of NHC in plasma: Treatment D versus Treatment A | Pre-dose, and at designated timepoints up to 72 hours postdose
  CL/F of NHC in plasma will be determined.
Vz/F of NHC in plasma: Treatment D versus Treatment A | Pre-dose, and at designated timepoints up to 72 hours postdose
  Vz/F of NHC in plasma will be determined.
Number of participants who experience one or more adverse events (AEs) | Up to ~ 38 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study intervention due to an AE | Up to ~ 38 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- QPS-MRA, LLC-Early Phase (Site 0002), South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Fiore JL, Jin Y, Heimbach T, Patel SR, Zhao T, Matthews CZ, Pagnussat S, Maas BM, Cheng MH, Stoch SA. Pharmacokinetics and bioequivalence of a molnupiravir tablet formulation compared with the molnupiravir capsule formulation in healthy adult participants-a randomized, open-label, three-period, crossover study. Antimicrob Agents Chemother. 2025 Mar 5;69(3):e0143424. doi: 10.1128/aac.01434-24. Epub 2025 Feb 6. PMID 39912659
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com